CLINICAL TRIAL: NCT03620617
Title: Beneficial Effects of Raspberry in Overweight/Obese Individuals: Potential Role of the Gut Microbiota in Alleviating the Metabolic Syndrome
Brief Title: Effect of Raspberry on Gut Microbiota and Metabolic Syndrome
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Responsible Party: Principal Investigator, Marie-Claude Vohl, Professor, Laval University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: RAMI 2017-218
Record Dates: First submitted 2018-08-01; First posted 2018-08-08 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Gut Microbiota; Metabolic Syndrome
Keywords: Raspberry; Diet
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Raspberry supplementation (Experimental): Dietary Supplement: 280g of frozen raspberries, taken daily for 8 weeks. Subjects will consume frozen raspberry to test if there is a significant difference on the impact on gut microbiota composition and metabolic syndrome parameters between this treatment and control group (without raspberry).
  Interventions: Dietary Supplement: Raspberry supplement
- Control (No Intervention): Control: follow their usual diet (control group). Subjects will follow their usual diet and not consume raspberry to test if there is a significant difference on the impact on gut microbiota composition and metabolic syndrome parameters between this treatment and the experimental group (with raspberry).

INTERVENTIONS:
Dietary Supplement: Raspberry supplement — During the 8-week protocol, participants will be invited either to consume 280g of frozen raspberries daily (morning and evening). The daily dose is equivalent to 2 cups of raspberries.
  Arms: Experimental: Raspberry supplementation

SUMMARY:
There is growing evidence that nutritional intervention with dietary polyphenols can positively modulate the gut microbiota to improve cardiometabolic health. Whether the beneficial effects of raspberry on obesity and the metabolic syndrome can be linked to their potential impact on the gut microbiota and intestinal integrity remains speculative at this time. Moreover, the mechanisms of action underlying health benefits associated to raspberry consumption are still unknown. The investigators are thus proposing to combine the study of metagenomics, transcriptomics and metabolomics to test whether a prebiotic activity of raspberry can play a role in the prevention of obesity-linked metabolic syndrome in a clinical setting.

ELIGIBILITY:
Inclusion Criteria:

* Men and premenopause women in good health
* Caucasians
* At least one of the following : BMI between 25 and 40 kg/m2 or Waist circumference ≥ 80 cm for women and ≥ 94 cm for men
* At least one of the following : TG ≥ 1.35 mmol/L or fasting insulinemia ≥ 42 pmol/L

Exclusion Criteria:

* Metabolic disorders (hypertension, diabetes, hypercholesterolemia)
* Regular use of medication affecting study parameters
* Use of natural health product in the last 3 months
* Use of antibiotics in the last 3 months
* Nicotine users
* Allergy or intolerance for raspberries
* Raspberry taste aversion
* More than 2 alcohol drinks par day
* Particular dietary habits (vegetarism, gluten-free diet, cetogenic diet...)
* Weight change of more than 5% in the last 3 months
* Surgery in the last 3 months or planed during the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2018-01-08 (Actual); Primary Completion 2019-08-22 (Actual); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Changes in plasma insulin/glucose of overweight/obese men and women taking frozen raspberries daily or following their usual diet (control group). | 12 months
Changes in plasma lipides/lipoproteins of overweight/obese men and women taking frozen raspberries daily or following their usual diet (control group). | 12 months

SECONDARY OUTCOMES:
Changes in gene expression in overweight/obese men and women taking frozen raspberries daily or following their usual diet (control group). | 3-6 months
Changes in metabolites concentration in overweight/obese men and women taking frozen raspberries daily or following their usual diet (control group). | 3-6 months
Changes in the gut microbiota composition in overweight/obese men and women taking frozen raspberries daily or following their usual diet (control group). | 3-6 months
Changes in systolic and diastolic blood pressure of overweight/obese men and women taking frozen raspberries daily or following their usual diet (control group). | 12 months
Changes in intestinal integrity (plasma lipopolysaccharide (LPS) and LPS binding protein (LBP) will be measured) of overweight/obese men and women taking frozen raspberries daily or following their usual diet (control group). | 12 months
Changes in inflammation biomarkers of overweight/obese men and women taking frozen raspberries daily or following their usual diet (control group). | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Claude Vohl, Principal Investigator — Laval University
Locations (1):
- Laval University, Québec, Canada

REFERENCES:
- [Derived] Franck M, de Toro-Martin J, Varin TV, Garneau V, Pilon G, Roy D, Couture P, Couillard C, Marette A, Vohl MC. Raspberry consumption: identification of distinct immune-metabolic response profiles by whole blood transcriptome profiling. J Nutr Biochem. 2022 Mar;101:108946. doi: 10.1016/j.jnutbio.2022.108946. Epub 2022 Jan 10. PMID 35016998